CLINICAL TRIAL: NCT04960592
Title: Epigenetic Mechanisms and Symptom Clusters Associated with the Resolution of Persistent Pain Following Spinal Cord Stimulation
Brief Title: Epigenetic Mechanisms and Symptom Clusters Associated with Resolution of Pain Following Spinal Cord Stimulation
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 260886
Record Dates: First submitted 2021-06-28; First posted 2021-07-14 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Stimulation; Chronic Pain
Keywords: SCS; Epigenetic; Persistent Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood samples will be drawn at Baseline visit, 90 day post baseline visit, and approximately 1 year post procedure follow up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SCS Responders: Patients who receive Spinal Cord Stimulation treatment and experience greater than 50% reduction in pain score following treatment.
  Interventions: Device: Spinal Cord Stimulation
- SCS Non Responders: Patients who receive Spinal Cord Stimulation treatment and do not experience greater than 50% reduction in pain score following treatment.
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Temporary implantation of a clinical available neurostimulator.

SUMMARY:
Spinal cord stimulation (SCS) is indicated for selected patients with chronic pain who have not responded to conventional medical management.

Forty (40) patients indicated for SCS placement and presenting to the University of Arkansas for Medical Sciences (UAMS) Interventional Pain Management Clinic in Little Rock, Arkansas will be recruited for this study. Prior to temporary stimulator placement, patients will complete symptom-related questionnaires and provide a blood sample. Demographic and clinical characteristics will be obtained through medical record review. Patients will complete the same questionnaires and provide a blood sample at each of the routine clinical care follow-up visits.

DETAILED DESCRIPTION:
Neuromodulation has emerged as a minimally invasive therapy effective for the treatment of refractory neuropathic pain conditions. Epidural placement of electrodes provides long term analgesia through electrical stimulation of the spinal cord which alters expression of genes involved in synaptic signaling in the dorsal horn. Patients who receive SCS represent a unique opportunity to study the physiological mechanisms associated with the resolution of chronic pain.

This is a descriptive, prospective, longitudinal study that will consist of individuals with persistent pain and meet criteria for implantation of a neurostimulation device. One hundred patients indicated for neurostimulation device placement and presenting to the University of Arkansas for Medical Sciences Interventional Pain Management Clinic in Little Rock, Arkansas will be recruited for this study. Patients who meet study inclusion criteria will be recruited to participate prior to stimulator placement procedure. Following an initial consultation and exam by a physician, patients will have necessary imaging and neuropsychological evaluation. Prior to SCS placement procedure, the patient will complete preoperative labs.

At baseline, patients will be asked to complete the demographic questionnaire, and physical functioning questionnaires, and provide a blood sample. Blood samples will be drawn and stored until sample processing is completed. Medical records will be reviewed and abstracted for research-related data elements from electronic medical records. Questionnaire and form responses are collected and recorded for study use.

Study time points for data collection and sample collection are Baseline (Pre-treatment), routine follow-up visit < 60 days after baseline, 3 months, and 1-year post-implant procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age greater than or equal to18 years) who meet clinical criteria for implantation of a neuromodulation device
* Able to speak, write, and understand English

Exclusion Criteria:

* Evidence of monetary gain related to the outcome of the procedure (example worker's compensation, ongoing litigation, pending disability claim)
* Pain greater than 4/10 on pain scale at a bodily site not being treated by the neuromodulation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the UAMS Interventional Pain Management Clinic and Neurosurgery Clinic indicated for a trial neuromodulator device placement. Potentially eligible patients will be identified by health care providers during routine clinic visits. Target enrollment is 100 participants for this study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Genes and regulatory regions associated with the resolution of chronic pain | 24 months
  Identification of genes that are associated with the resolution of pain
Changes in the day to day functioning | 24 months
  Identification of psychosocial measures (i.e., patient reported outcome measures; pain catastrophizing) and patient reported functioning associated with the resolution of pain

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Stephens, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
The PI will monitor study procedures to protect the safety of research subjects, the quality of the data and the integrity of the study. Results of this study may be used for presentations, posters, or publications. The publications will not contain any identifiable information that could be linked to a participant. The final, anonymized dataset will be made publicly available upon publication of study findings.